CLINICAL TRIAL: NCT07350980
Title: The Effect of Scents Applied During Heel Blood Collection on Newborn Crying Duration, Pain, and Physiological Parameters; A Randomized Controlled Study.
Brief Title: The Effect of Scents Applied During Heel Blood Collection on Newborn Crying Duration, Pain, and Physiological Parameters
Acronym: Randomized
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, öznur tiryaki, Associate Professor, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Oznur T.
Record Dates: First submitted 2025-12-28; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Neonatal; Pain Management
Keywords: newborn
MeSH Terms: conditions — Agnosia | interventions — Oils

STUDY DESIGN:
Intervention Model Description: 2 intervention, 1 control
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intervention group (Lavender) (Experimental): Lavender
  Interventions: Other: oil
- intervention group (tangerine) (Experimental): tangerine
  Interventions: Other: oil
- Control group (No Intervention): rutin

INTERVENTIONS:
Other: oil — experiment
  Arms: intervention group (Lavender); intervention group (tangerine)

SUMMARY:
One of the most common and painful procedures in newborns is taking a capillary blood sample from the heel. This basic procedure, widely used in early health assessments, particularly in newborn screening tests, can cause mild to moderate pain.While both pharmacological and non-pharmacological approaches are used in pain management in newborns, the primary goal is to minimize and prevent painful stimuli as much as possible. Non-pharmacological methods are preferred in newborn care because they have no side effects, are easy to apply, low-cost, and caregiver-friendly.

DETAILED DESCRIPTION:
This study was designed as a prospective, three-arm, parallel-group randomized controlled trial. It focused on non-pharmacological methods (lavender oil, mandarin oil, control group/standard care).Mothers of newborns meeting the recruitment criteria were informed of the study before heel prick testing and provided verbal and written consent. The standard approach involves performing heel prick testing on all newborns in their mothers' arms.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 38-42 weeks,
* APGAR score of 7 or higher at 5 minutes,
* Neither mother nor baby should have used sedatives, tranquilizers, or anticonvulsants in the last 24 hours,
* Heel prick blood should be planned as part of the routine neonatal screening program,
* No blood should be taken from the heel prick for any other reason before the procedure,
* Parents should voluntarily participate in the study.

Exclusion Criteria:

* Gestational age of 37 weeks or less,
* APGAR score of 6 or lower at 5 minutes,
* Having a diagnosed lung disease,
* Having a history of atopic dermatitis, hypersensitivity, or allergies,
* Parents should not wish to participate in the study.

Ages: 37 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2025-06-25 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
crying times | Before the procedure, during the procedure, and for a total of 10 minutes after the procedure.
  measuring the crying duration with a stopwatch
heart rate | Before the procedure, during the procedure, and for a total of 10 minutes after the procedure.
  Measurement with pulse oximeter
Neonatal infant pain scale | Before the procedure, during the procedure, and for a total of 10 minutes after the procedure.
  The scale includes f ive behavioral parameters (facial expression, crying, armmovements, leg movements, and state of arousal) and one physiological parameter (breathing patterns). Each behavior is scored 0-1; the crying parameter is scored 0-1-2. The lowest score is 0 and the highest score is 7.

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Ethically, patient information can be shared upon reasonable request without revealing their identities for security reasons